CLINICAL TRIAL: NCT01551472
Title: Prospective Multicenter Open Label Study Examining the Mid- and Long-term Safety and Efficacy of the 3DKnee™ System With Vitamin E UHMWPE Tibial Inserts (3DKnee™ With E-plus Insert)
Brief Title: Post Market Study of the 3DKnee™ With E-plus Insert
Acronym: e-plus
Status: Terminated | Type: Observational
Why Stopped: Lack of sufficient enrollment
Sponsor: Encore Medical, L.P. (Industry)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: PS-706
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Degenerative Joint Disease; Osteoarthritis; Traumatic Arthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3DKnee™ with e-plus Insert: Subjects who meet the indications for use criteria for the 3DKnee™ System with vitamin E UHMWPE tibial inserts (VE) and who are candidates for a primary knee arthroplasty.
  Interventions: Device: 3DKnee™ System with Vitamin E UHMWPE Tibial Inserts

INTERVENTIONS:
Device: 3DKnee™ System with Vitamin E UHMWPE Tibial Inserts — This device is part of a total knee replacement system utilized in treating patients who are candidates for primary cemented total knee arthroplasty or revision arthroplasty where bone loss is minimal and the collateral ligaments are intact. It is intended to aid the surgeon in relieving the patient of knee pain and restoring knee joint function.

SUMMARY:
The purpose of this study is to evaluate the use and efficacy of the 3DKnee™ System using Vitamin E UHMWPE tibial inserts for total knee replacement surgery.

DETAILED DESCRIPTION:
Total knee replacement surgery is widely accepted as effective treatment for degenerative joint disease (DJD), osteoarthritis and rheumatoid arthritis. Relief of patient pain and return of mobility are the primary goals that can be accomplished by this surgery. Currently available prosthetic designs accomplish these goals and the surgery has been defined as one of the most successful operations available to improve the quality of life for patients with DJD. This study will evaluate subjects who are candidates for a total knee replacement and meet the indications for use criteria for the 3DKnee™ System with vitamin E UHMWPE tibial inserts (VE).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for a total primary knee replacement.
* Subject must have knee joint disease related to degenerative joint disease, including osteoarthritis or traumatic arthritis
* Subject has a BMI ≤ 40.00 kg/m2
* Subject is likely to be available for evaluation for the duration of the study
* Subject is able and willing to sign the informed consent and follow study procedures
* Subject is not pregnant
* Subject must be between age 40 and age 75 at the time of consent

Exclusion Criteria:

* Subject has had a prior total or uni-knee replacement on this knee in the past (no revisions allowed in study)
* Subject has avascular necrosis of the femoral condyles, post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy, moderate valgus, varus, or flexion deformities or rheumatoid arthritis
* Subject has an active cancer or is a survivor for <5 years except for squamous cell or basal cell skin cancer
* Subject has a chronic disease(s) where, in the opinion of the investigator, the disease will interfere with the patient's ability to follow the protocol
* Subject is currently a documented substance abuser (alcohol or other addictions)
* Subject has an infection, or history of infection (within the last 3 months), acute or chronic, local or systemic
* Subject has a history of muscular, neurological or vascular deficiencies which compromise the affected extremity
* Subject has a BMI > 40.00 kg/m2
* Subject has loss of ligamentous structures
* Subject has high levels of physical activity and is unwilling to modify levels of physical activity commensurate with recommendations
* Subject has a mental condition that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject is a prisoner
* Subject is pregnant
* Subject has known materials sensitivity (to metals)
* Subject is younger than 40 years (<40) or older than 75 years (>75) at the time of consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must be diagnosed with either osteoarthritis or traumatic arthritis and be candidates for a primary total knee arthroplasty. They must also meet the indications for use for the 3DKnee system with the vitamin E tibial insert.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of the Vitamin E UHMWPE as part of the total knee system, measured by Knee Society Score Evaluation and total number of radiologic failures of the device. | 2 year
  The (American) Knee Society Score has both an objective and a functional component. The objective score takes into account pain, flexion, stability, alignment, extension lag and flexion contracture. Overall success will be defined as a KSS score ≥ 80 at two years.
  Radiolucencies have been defined as two types, with one type being more common than the other. In the case of physiologic radiolucency, which is the most common type of radiolucency seen, there is a narrow line present that is well-defined around the prosthesis. This line is surrounded by a radio-dense line and tends to consolidate (disappear) within the first year. The second type of radiolucency, the pathologic radiolucency, is rarer and is associated with loosening and infection. It is a progressive, poorly defined radiolucency that is more than 2 mm thick and without a radiolucent line.

SECONDARY OUTCOMES:
Change in Knee Society Score from pre-surgery to 10 years | 10 year
  The Knee Society Score includes a knee rating and function score. This evaluation covers the knee rating score with three main parameters of pain, stability and range of motion and that flexion contracture, extension lag and misalignment should be dealt with as deductions. Thus, 100 points will be obtained by a well-aligned knee with no pain, 125 degrees of motion, and negligible anteroposterior and mediolateral instability. 50 points are allotted for pain, 25 for stability, and 25 for range of motion. Grading for KS Score: Excellent (90-100), Good (80-90), Fair (70-79) and Poor (<70).
Change in WOMAC Osteoarthritis Index from pre-surgery to 10 years | 10 year
  The Western Ontario McMaster Arthritis Index is a set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip. It can be self-administered. It assesses the pain, joint stiffness, physical, social & emotional function of a person with osteoarthritis in determining the overall level of disability.
Change in Oxford Knee Score from pre-surgery to 10 years | 10 year
  The Oxford Knee Score (OKS) is a patient-based outcomes measure consisting of 12 questions that is sensitive, simple and validated. It is based on a maximum score of 48.
Change in response to Quality of Life questions from pre-surgery to 6 months and each year thereafter through 10 years | 10 years
6. Change in pain from pre-surgery to 6 months and each year thereafter through 10 years | 10 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Orthopaedic Surgery Specialists, Burbank, California
  - Orthopedic Specialists of North County, Oceanside, California
  - Institute for Orthopaedic Surgery and Sports Medicine, Fort Myers, Florida
  - St. Peter's Bone & Joint Surgery, City of Saint Peters, Missouri
  - New Mexico Orthopedics, Albuquerque, New Mexico
  - Texas Institute for Hip and Knee Surgery, Austin, Texas